CLINICAL TRIAL: NCT03754374
Title: Health Care Access for Asylum Seekers in Brittany : Description, Associated Factors and Levers of Improvement
Acronym: ACCEDAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_9852_ACCEDAB
Record Dates: First submitted 2018-11-22; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Adult Asylum Seekers Who Have Applied for Asylum at the Regional Prefecture in Rennes
Keywords: Primary health; migrants; health care utilization; access to healthcare
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: access to healthcare — use or non-use of dedicated health facilities

SUMMARY:
The main objective of this research is to study the logics and the associated factors with asylum seekers use of dedicated health structures.

This objective aims to address major concerns related to the entry and continued participation in the health care system of asylum seekers, including the medical and social dimensions.

It aims to produce, then analyze and disseminate data on the factors associated with seeking asylum seekers to optimize the care of migrants in the French health system

ELIGIBILITY:
Inclusion Criteria:

- Adult asylum seekers who have applied for asylum in the prefecture of Brittany from May 22, 2018 to May 21, 2019 (or one year after obtaining authorization from the CCTIRS and the CNIL).

Exclusion Criteria:

* Migrants not asylum seekers (with tourist visa, migrants of the European Union (foreign nationality and not membership in the Schengen area), migrants arriving in a family reunification, migrant in irregular situation).
* Minor : unaccompanied foreign minor or with their family
* Incapacity of a person to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult asylum seekers who have applied for asylum in the prefecture of Brittany
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2019-11-22 (Estimated)

PRIMARY OUTCOMES:
Use of health care structure | 6 months
  Factors associated with the use or non-use of dedicated health facilities will be the individual (sociodemographic, migration), organizational (access to rights, characteristics of the organization of dedicated structures) and the environment characteristics reported by asylum seekers having or not having recourse to the dedicated health structures.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Jarno, MD, Principal Investigator — Rennes University Hospital
Locations (2):
- France (2):
  - COALLIA - Plateforme d'accueil des demandeurs d'asile, Rennes
  - CHU de Rennes, Rennes